CLINICAL TRIAL: NCT03952455
Title: Deep Brain Stimulation of the Bilateral Nucleus Accumbens for Patients With Methadone Maintenance Treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Bomin Sun, Director of the Department of Functional Neurosurgery, Ruijin Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019 NAc-DBS MMT
Record Dates: First submitted 2019-05-14; First posted 2019-05-16 (Actual); Last update posted 2020-01-10 (Actual); Status verified 2019-05

CONDITIONS: Addiction Opiate
Keywords: Nucleus Accumbens; Deep brain stimulation; Methadone
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DBS (Experimental): All subjects will undergo bilateral surgical implantation of DBS system in the Nucleus Accumbens. The DBS system will be active at two days after surgery.
  Interventions: Procedure: Bilateral surgical implantation of DBS system to Nucleus Accumbens

INTERVENTIONS:
Procedure: Bilateral surgical implantation of DBS system to Nucleus Accumbens — We plan to use the SceneRay 1242 (SceneRay, SuZhou, China) electrode with a diameter of 1.27 mm and 4 contacts. The SceneRay 1242 electrode combined with the SceneRay 1181 implantable pulse generator has the advantage of adaptive coverage area for the Ventral Capsule/Ventral Striatum, enabling simultaneous implantation in the nucleus accumbens (NAc; 2 ventral contacts) and the anterior limb of the internal capsule (ALIC; 2 dorsal contacts) with independently programmed parameters such as frequency, amplitude, and voltage; and remote and wireless programing, which allows for convenient and prompt adjustments in emergency situations. The contact length is 3.0 mm and the spacings between the ventral and dorsal contacts are 2 mm, 4 mm, and 4 mm, respectively, spanning a total length of 22.5 mm (3 + 2 + 3 + 4 + 3 + 4 + 3 mm, with 0.5 mm projecting from the electrode tip).

SUMMARY:
Methadone maintenance treatment (MMT) is one of the main forms of treatments for opioid dependence. Despite its effectiveness and widespread use, people will experience withdrawal if daily dose is insufficient or missed, promoting reluctance to attempt detoxification. In addition, methadone is a full opioid agonist which can induce respiratory depression or sedation without ceiling level, so overdose usage can be fatal. Hence, an alternative therapy is needed to completely reduce the carving for drugs and to relieve the negative affective sate caused by withdrawal.

Deep brain stimulation (DBS) is a reasonable treatment approach for addiction. Since 2009 the first case report emerged, the nucleus accumbens (NAc) is still the only brain target to be investigated in clinical case series of DBS for alcohol and heroin addiction.

This research will mainly investigate the effectiveness and safety of NAc-DBS for patients with methadone maintenance treatment. The investigators will also explore the influence of NAc-DBS on brain activity and cognition.

ELIGIBILITY:
Inclusion Criteria:

* MINI diagnosis of substance dependence;
* Proficiency in Mandarin language;
* Failure to detox more than three times;
* Long-term methadone maintenance treatment;
* Capacity to provide informed consent (understanding of the study purpose and methods);

Exclusion Criteria:

* Schizophrenia(MINI diagnosis);
* Antisocial personality disorder(MINI diagnosis);
* Contraindications of a MRI-examination, e.g. implanted cardiac pacemaker/heart defibrillator;
* Severe cognitive impairments(MoCA ≤ 22);
* Enrollment in other clinical trials;
* Stereotactic respectively neurosurgical intervention in the past;
* Contraindications of stereotactic intervention, e.g. increased bleeding disposition, cerebrovascular diseases (e.g. arteriovenous malfunction, aneurysms, systemic vascular diseases);
* Serious or instable organic diseases (e.g. instable coronal heart disease);
* Tested positively for HIV;
* Pregnancy and/or lactation;
* Epilepsy or other severe brain trauma or neurological impairments;

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2019-05-13 (Actual); Primary Completion 2021-06-01 (Estimated); Study Completion 2021-06-01 (Estimated)

PRIMARY OUTCOMES:
Changes in Methadone dose | Baseline (preoperative),1 month, 3 months,6 months,9 months, 12 months
  The volume of daily methadone the patients used.

SECONDARY OUTCOMES:
Hamilton Depression Scale(HAMD-17) | Baseline(preoperative),1 month, 3 months, 6 months, 9 months, 12 months
  17 items, Total scores<7: normal; 7<Total scores≤17: possible depression; 17<Total scores≤24: definite depression; Total score>24: severe depression
Hamilton Anxiety Scale (HAMA) | Baseline(preoperative),1 month, 3 months, 6 months,9 months, 12 months
  14 items, Total scores<6: normal; 7<Total scores≤14: possible anxiety; 14<Total scores≤21:definite anxiety; Total score>21: severe anxiety
Young Manic Rating Scale (YMRS) | Baseline(preoperative),1 month, 3 months, 6 months,9 months, 12 months
  The Young Mania Rating Scale (YMRS) is one of the most frequently utilized rating scales to assess manic symptoms. The scale has 11 items and is based on the patient's subjective report of his or her clinical condition.
Monitoring of Side Effects Scale (MOSES) | Baseline(preoperative),1 month, 3 months, 6 months,9 months, 12 months
  To evaluate side effects. The higher score means more severity of side effects.
Changes in Subjective Opiate Withdrawal Scale(SOWS) | Baseline(preoperative),1 month, 3 months, 6 months,9 months, 12 months
  Subjective Opiate Withdrawal Scale is a 16-item self-reported scale assessing severity of opiate withdrawal. Each item is rated on a 5-point Likert scale, ranging form 0(not at all) to 4(extremely).
Obsessive compulsive drug use scale(OCDUS) | Baseline(preoperative),1 month, 3 months, 6 months,9 months, 12 months
  Obsessive compulsive drug use scale is a 13-item self-rating scale measuring opiate craving. The total score ranges from 0 to 52. The higher score indicates stronger carving.
The MOS item short from health survey (SF-36) | Baseline(preoperative),1 month, 3 months,6 months,9 months, 12 months
  36 items. To evaluate the quality of life and the higher score indicates better quality of life.
World Health Organization Quality of Life-BREF (WHO-BREF) | Baseline(preoperative),1 month, 3 months,6 months,9 months, 12 months
  26 items. The higher score means the better quality of life.
Fagerstrom Test for Nicotine Dependence assessment (FTND) | Baseline(preoperative),1 month, 3months,6months,9 months, 12 months
  To evaluate Nicotine Dependence. The higher of scores indicates higher level of Nicotine Dependence
Beck depression inventory(BDI) | Baseline(preoperative),1 month, 3months,6months,9 months, 12 months
  The BDI contains 21 questions, each answer scored on a scale value of 0 to 3. 0-13: minimal depression;14-19:mild depression; 20-28:moderate depression; and 29-63:severe depression. Higher total score indicate more severe depressive symptoms.
Beck anxiety inventory(BAI) | Baseline(preoperative),1 month, 3months,6months,9 months, 12 months
  The BAI contains 21 questions, each answer scored on a scale value of 0 to 3. 0-21: mild anxiety;22-35: moderate anxiety;36-63:severe anxiety. Higher total score indicate more severe anxiety symptoms.
Perceived stress scale(PSS-10) | Baseline(preoperative),1 month, 3months,6months,9 months, 12 months
  The PSS-10 is a classic stress assessment instrument. Each item is rated on a 5-likert scale ranging form 0(never) to 4(often). Higher score indicate more severity of stress symptom.
Twenty Item Positive and Negative Affect Schedule (PANAS) | Baseline(preoperative),1 month, 3months,6months,9 months, 12 months
  The PANAS contains two subscales: positive and negative subscale. Each item is rated on a 5-likert scale ranging from 1(Not at all) to 5(severely, it bothered me a lot).
Work and Social Adjustment Scale(WSAS) | Baseline(preoperative),1 month, 3months,6months,9 months, 12 months
  Self-rated scale. The maximum score of the WSAS is 40, lower scores are better.
Cognitive performance | Baseline(preoperative),6 months,12 months
  Cognitive performance is measured by a series of tasks which include stop signal task, paired associated memory, spatial working memory, stocking of Cambridge, intra-extra dimensional set shift, Bart, Beads, Delay discounting task, model-based and model-free task, avoid-approach task, dot-probe task, drug rating task.
Brain activity | Baseline(preoperative), 6 months,12 months
  PET(Positron Emission Tomography) or fMRI(functional Magnetic Resonance Imaging) are used in this study.

OTHER OUTCOMES:
Barratt impulsiveness scale | Baseline(preoperative)
  The Barratt Impulsiveness Scale is a questionnaire designed to assess the personality/behavioral construct of impulsiveness which is composed of 30 items describing common impulsive or non-impulsive (for reverse scored items) behaviors and preferences. It has three 2nd order facets which are attentional, motor and non-planning. Each facet has 10 items. Higher score means greater impulsivity.
UPPS-P impulsive behavior scale | Baseline(preoperative)
  The UPPS-P Impulsive Behavior Scale is a 59-item questionnaire assessing impulsive personality traits. Each item is rated on a 4-point scale ranging from 1 (agree strongly) to 4 (disagree strongly) to indicate subject's agreement with statements. This scale includes the following five subscales: negative urgency (NU), lack of premeditation (LPM), lack of perseverance (LPS), sensation seeking (SS) and positive urgency (PU). Higher score represents a greater level of impulsivity.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Ruijin Hospital Functional Neurosurgery, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Background] Muller UJ, Voges J, Steiner J, Galazky I, Heinze HJ, Moller M, Pisapia J, Halpern C, Caplan A, Bogerts B, Kuhn J. Deep brain stimulation of the nucleus accumbens for the treatment of addiction. Ann N Y Acad Sci. 2013 Apr;1282:119-28. doi: 10.1111/j.1749-6632.2012.06834.x. Epub 2012 Dec 10. PMID 23227826
- [Background] Kuhn J, Moller M, Treppmann JF, Bartsch C, Lenartz D, Gruendler TO, Maarouf M, Brosig A, Barnikol UB, Klosterkotter J, Sturm V. Deep brain stimulation of the nucleus accumbens and its usefulness in severe opioid addiction. Mol Psychiatry. 2014 Feb;19(2):145-6. doi: 10.1038/mp.2012.196. Epub 2013 Jan 22. No abstract available. PMID 23337942
- [Background] Muller UJ, Sturm V, Voges J, Heinze HJ, Galazky I, Buntjen L, Heldmann M, Frodl T, Steiner J, Bogerts B. Nucleus Accumbens Deep Brain Stimulation for Alcohol Addiction - Safety and Clinical Long-term Results of a Pilot Trial. Pharmacopsychiatry. 2016 Jul;49(4):170-3. doi: 10.1055/s-0042-104507. Epub 2016 May 4. PMID 27145161